CLINICAL TRIAL: NCT05765695
Title: Radiofrequency Ablation for Treating Thyroid Nodules Classified as TIR3A, With a Negative Genetic Evaluation for Thyroid Carcinoma
Brief Title: Radiofrequency Ablation in TIR3A Nodules With Negative Genetic Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05C023
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Nodule
Keywords: thyroid nodule; indeterminate; genetic; radiofrequency ablation; follow-up
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated group (Experimental)
  Interventions: Procedure: Radiofrequency ablation performed with a 19 gauge STARmed needle.

INTERVENTIONS:
Procedure: Radiofrequency ablation performed with a 19 gauge STARmed needle. — The ablation with radiofrequency is a safe and effective minimally invasive procedure that results in thermal tissue necrosis. A needle electrode is inserted into the thyroid nodule using ultrasound guidance and generates heat by alternating electric current causing thermal injury. Afterwards, the ablated tissue is gradually absorbed with progressive shrinkage of the nodule.

SUMMARY:
The goal of this clinical trial is to demonstrate that TIR3A nodules with negative genetic test can be safely and effectively treated by radiofrequency ablation, with nodular shrinkage and improvement of clinical symptoms.

Fine needle aspiration cytology is the gold standard test for differential diagnosis of thyroid nodules, but sometimes the result can be indeterminate with a risk of malignancy of 10-30%. In these cases the ablation is not indicated and many patients with benign nodules that may benefit from the procedure are not treated.

All the patients enrolled must have a TIR3A cytology and negative genetic test for mutations associated with thyroid carcinoma. Before the ablation blood, evaluation of serum TSH, anti-thyroglobulin antibodies, anti-thyroid peroxidase antibodies and calcitonin levels will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thyroid nodule eligible for radiofrequency ablation, with low-risk indeterminate lesion cytology (TIR3A) and negative genetic test for mutations associated with thyroid carcinoma

Exclusion Criteria:

* Patients who are not able to sign the informed consent
* Patients with contraindications to radiofrequency ablation
* Patients with cytology different from TIR3A
* Patients with positive genetic test for mutations associated with thyroid carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Thyroid nodule volume reduction rate | 1 month after the procedure
  The change rate of the thyroid nodule volume after radiofrequency ablation compared to baseline
Thyroid nodule volume reduction rate | 6 months after the procedure
  The change rate of the thyroid nodule volume after radiofrequency ablation compared to baseline
Thyroid nodule volume reduction rate | 12 months after the procedure
  The change rate of the thyroid nodule volume after radiofrequency ablation compared to baseline
Complication rate | When the procedure is performed
  Assessment of the complications of the procedure and over time
Complication rate | 1 month after the procedure
  Assessment of the complications of the procedure and over time
Complication rate | 6 months after the procedure
  Assessment of the complications of the procedure and over time
Complication rate | 12 months after the procedure
  Assessment of the complications of the procedure and over time

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy